CLINICAL TRIAL: NCT01571752
Title: Health Outcomes by Neighborhood - HON Study Baltimore
Brief Title: Health Outcomes by Neighborhood - Baltimore
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912472; 12-DA-N472
Record Dates: First submitted 2012-04-04; First posted 2012-04-05 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-04

CONDITIONS: Stigma; Activity Space; Social Networks; HIV Status; Drug Abuse/Dependence
Keywords: Drug Abuse; Ecological Momentary Assessment (EMA); Environment; Genetic; Longitudinal; Natural History
MeSH Terms: conditions — Social Stigma; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- CMU: Current marijuana users
- Cohort 1 - NIH Negative: HIV negative adults
- Cohort 1- HIV Positive: HIV positive adults
- Cohort 2 Seeds-Wave 0: HIV positive adults
- Cohort 2 Wave 1: HIV negative adults or HIV positive adults
- Cohort 2 Wave 2: HIV negative adults or HIV positive adults
- COSU: Current opioid/stimulant users
- COSU-NTS: Non-treatment seekers
- COSU-TS: Treatment seekers
- NDU: Non-drug-users
- Unclassified

SUMMARY:
Background:

- Researchers have been studying patterns of mood and drug use in specific neighborhoods. This study will look at environmental factors that may affect drug use, addiction, and treatment seeking in Baltimore neighborhoods. The results could inform prevention efforts, enhance treatment interventions, and improve substance use outcomes.

Objectives:

- To better understand why some people start to use drugs, why some people who use drugs become addicted, and why some people who become addicted enter treatment.

Eligibility:

- Individuals at least 18 years of age who are living in the neighborhoods participating in the study.

Design:

* Participants will be screened with a physical exam and medical history. They will be separated into one of four groups: (1) people who do not use drugs, (2) people who have used drugs in the past, (3) people who are using drugs and want treatment, and (4) people who are using drugs and do not want treatment.
* This study will include two outpatient visits about 12 months apart. Each visit will last about 5 hours. Each study visit may be done in 1 day or in 2 days.
* At each study visit, participants will provide blood, breath, urine, and saliva samples. They will also have a heart function test and body measurements. They will complete questionnaires about personal and family history.
* There will be monthly follow-up phone calls between the two visits.

DETAILED DESCRIPTION:
Phase B

Background. The reasons for initiation and continuation of use of illicit substances are multifactorial; however, some individuals appear resistant to both. One set of determinants lies in the environment. In ongoing studies, we are examining environmental concomitants of behavior in individuals in drug treatment. In this study, we will examine environmental factors that may impact initiation, addiction, and treatment seeking among the greater population at large (nondrug-users, current opioid/stimulant users, and current marijuana users).

Scientific goals. (1) To assess, cross-sectionally at baseline, differences in stress, social stability, and mental and physical health among three main neighborhood-matched groups of current opioid/stimulant users, current marijuana users, and nondrug users; (2) to assess, longitudinally, mediators of 12-month changes in drug-misuse status in the same three groups; (3) to provide neighborhood-matched control groups of non-drug-using individuals, Unclassified/former drug users, and current opioid/stimulant drug users not seeking treatment for our ongoing environmental studies of individuals in drug treatment; (4) to explore the possible role of genetics and its interplay with environment in regards to drug use initiation, addiction, and treatment seeking among the study groups, (5) to assess EMA reports of drug use and psychosocial stress as well as real-time environmental risk exposure in a non-treatment seeking and/or nondrug using population and compare to our ongoing environmental studies of individuals in drug treatment, (6) to assess the accuracy of stress detection in the lab and the field by the Health Tag.

Participant population. We will enroll 650 participants in Phase B of the study for a total enrollment (Phase A + Phase B + Phase C) of 3000 participants. Target enrollment will include 25% women and 70% minorities (mostly African American).

Experimental design and methods. This is a three-group observational study with a crosssectional component and a longitudinal component: each participant will be assessed in two visits spaced approximately 12 months apart. For participants enrolled in Phase B after January 26, 2021, the interval between the two visits may be shorter than 12 months. The three main groups will be: (1) non-drug-users (NDUs), (2) current opioid/stimulant users [(COSUs) comprised of two subgroups: treatment seeking (COSU-TS) and non treatment seeking (COSU-NTS)], and current marijuana users (CMUs). All groups will be roughly matched for socioeconomic status and neighborhoods of residence. Each participant will attend a 3-5-hour initial study visit and a 3-5-hour 12 month visit #2. The study visits will include a questionnaire component and a biologicalsample component. Questionnaires will cover substance use, stress, social stability (including healthcare access/utilization, and neighborhood environment), physical and mental health (including quality of life, HIV, and trauma). The biological component will consist of samples of urine (for drugs of abuse and cotinine), breath (for alcohol and carbon monoxide). Blood for genetics will be obtained at Visit 1 or Visit 2. The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component). Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors. Individuals who choose not to return for a 12-month Visit #2 will be asked to complete a 45-minute telephone visit #2. For participants enrolled in Phase B after January 26, 2021, all participants will be asked to complete their visit #2 by telephone only. In the HON EMA/GMA secondary study participants will carry a smartphone for up to 4 weeks after completing Visit 1. Event-triggered entries will be initiated by participants (1) each time that they use a drug (COSU) or marijuana and/or alcohol (NDU, CMU, and Unclassified) and (2) each time they feel overwhelmed, anxious, or stressed more than usual. Participants will also make 5 random-signal-triggered recordings per day and one brief end of day recording. During this study participants will also complete compliance visits once per week. In the Health Tag secondary study, participants will undergo a one-day laboratory session followed by a 30-day field study. Benefits to participants and/or society. There are no benefits to participants. The knowledge gained may benefit society by providing data on the health outcomes of drug-using and non-drugusing individuals and the natural history of drug use by neighborhood.

Risks to participants. This is a minimal-risk study, consisting of standard physical and questionnaire-based assessments.

ELIGIBILITY:
* INCLUSION CRITERIA:

The enrollment target in Phase B is 650 community-dwelling individuals (at least 325 of whom we anticipate will provide 12-month Visit #2 data in our 3 main study groups). Enrollment for Phase A + Phase B + Phase C =3000.

* Age at least 18 years. Rationale: Children under 18 will not be included because many of the measures to be administered in this study are not validated for use with children. Furthermore, the research question under investigation is the drug trajectories of adults, over the age of 18. However, there is no intervention in this study that is contraindicated for older adults, and given that addiction in the elderly is understudied, it is important to include elderly individuals.
* Residence in Baltimore city or one of the surrounding counties. Rationale: Our current geographic mapping technology currently only includes these areas.

EXCLUSION CRITERIA:

-Inability to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll 650 participants in Phase B of the study for a total enrollment (Phase A + Phase B + Phase C) of 3000 participants. Target enrollment will include 25% women and 70% minorities (mostly African-American).
Sampling Method: Non-Probability Sample
Enrollment: 1651 (Actual)
Dates: Start 2012-07-17 (Actual)

PRIMARY OUTCOMES:
We will examine environmental factors that may impact initiation, addiction, and treatment seeking among the greater population at large (non-drug-users, current opioid/stimulant users, and current marijuana users) | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)
To provide neighborhood-matched control groups of non-drug-using individuals, Unclassified/former drug users, and current opioid/stimulant drug users not seeking treatment | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)
To explore the possible role of genetics and its interplay with environment in regards to drug use initiation, addiction, and treatment seeking among the study groups | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)
To assess, longitudinally, mediators of 12-month changes in drug-misuse status in the same three groups | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)
To assess the accuracy of stress detection in the lab and the field by the Health Tag | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)
To assess EMA reports of drug use and psychosocial stress as well as real-time environmental risk exposure in a non-treatment seeking and/or nondrug using population | 12 months
  The primary outcome measures will be lifetime substance-misuse history (cross-sectional component) and changes in drug-use status across the 12 months between visits (longitudinal component)

SECONDARY OUTCOMES:
Random-signal-triggered recordings | Daily
  Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors
One-day laboratory session | Once
  Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors
Clinic Compliance Visit | Weekly
  Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors
Brief end of day recording | Daily
  Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors
30-day field study | post-30 day
  Secondary outcome measures will include: biological assessments of drug use; medical, psychiatric, social determinants of health; and impulsivity and decision-making factors

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Leggio, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Panlilio LV, Preston KL, Bertz JW, Moran LM, Tyburski M, Hertzel SK, Husami S, Adan F, Epstein DH, Phillips KA. Objective Neighborhood-Level Disorder Versus Subjective Safety as Predictors of HIV Transmission Risk and Momentary Well-Being. AIDS Behav. 2024 Oct;28(10):3326-3337. doi: 10.1007/s10461-024-04413-z. Epub 2024 Jul 4. PMID 38965184
- [Derived] Moran LM, Panlilio LV, Hertzel SK, Bertz JW, Tyburski M, Etter JR, Epstein DH, Preston KL, Phillips KA. Health Outcomes by Neighborhood (HON): Effects of Neighborhood, Social Instability, and Health Factors on 12-Month Trajectories of Substance-Use Disorder Symptoms. Subst Use Misuse. 2023;58(12):1460-1472. doi: 10.1080/10826084.2023.2223258. Epub 2023 Jun 28. PMID 37380598
- [Derived] Stull SW, Panlilio LV, Moran LM, Schroeder JR, Bertz JW, Epstein DH, Preston KL, Phillips KA. The chippers, the quitters, and the highly symptomatic: A 12-month longitudinal study of DSM-5 opioid- and cocaine-use problems in a community sample. Addict Behav. 2019 Sep;96:183-191. doi: 10.1016/j.addbeh.2019.04.030. Epub 2019 Apr 29. PMID 31108264